CLINICAL TRIAL: NCT02747069
Title: Determination of Heart Rate in Neonates on the NICU and Delivery Suite Using ECG and Electronic Stethoscope, a Feasibility Study
Brief Title: HeartLight Pulse Study: Evaluation of Heart Rate Using an Electronic Stethoscope and Pre Placed ECG in the Delivery Room
Acronym: HLPulseS
Status: Suspended | Type: Observational
Why Stopped: New data available in public domain requires re-evaluation of protocol.
Sponsor: University of Nottingham (Other)
Collaborators: Heartlight Systems Limited (Industry)
Responsible Party: Sponsor
Other Study IDs: 15124
Record Dates: First submitted 2016-02-25; First posted 2016-04-21 (Estimated); Last update posted 2018-05-17 (Actual); Status verified 2018-05

CONDITIONS: Premature Birth
Keywords: Heart rate; Electronic Stethoscope; Electrocardiogram; Resuscitation
MeSH Terms: conditions — Premature Birth | interventions — Electrocardiography

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- NICU electronic stethoscope: Neonatal patients of any gestation admitted to the neonatal intensive care unit (NICU) and undergoing routine monitoring with ECG and pulse oximetry Heart rate will be evaluated using an electronic stethoscope
  Interventions: Device: NICU electronic stethoscope
- Newborns <32 weeks and ECG: Neonatal patients <32 weeks gestation Heart rate will be assessed at the time of delivery with both an electronic stethoscope and ECG using a pre placed lead system
  Interventions: Device: NICU electronic stethoscope; Device: Newborns <32 weeks and ECG

INTERVENTIONS:
Device: NICU electronic stethoscope — Assessment of heart rate using the electronic stethoscope for up to 10 minutes compared to ECG and pulse oximetry devices used to monitor neonates whilst on NICU
Device: Newborns <32 weeks and ECG — The three leads from the ECG device will be pre placed onto a plastic bag prior to delivery. The pre term infant (<32 weeks) placed into the bag at the time of delivery and heart rate will be assessed for up to 30 minutes
  Groups: Newborns <32 weeks and ECG

SUMMARY:
This study will evaluate the accuracy of both an electronic stethoscope and electrocardiogram (ECG) to evaluate heart rate in neonatal patients in the delivery suite.

The initial phase of this study will assess the electronic stethoscope use on stable neonates on the neonatal care prior to use in the delivery room.

DETAILED DESCRIPTION:
Up to 10% of newborns (79K/yr in United Kingdom, 13 million/yr worldwide) require some form of resuscitation at birth. It is estimated that approximately 7 million babies worldwide, especially the premature group, will require more advanced resuscitation. The correct, structured management of the resuscitation in the few 'golden' minutes after birth is critical to prevent significant morbidity (e.g. cerebral palsy due to asphyxiation) or death. There is strong evidence that standardised resuscitation training and algorithms significantly improve newborn outcomes and could reduce mortality by 30% in certain healthcare institution. International newborn resuscitation guidelines state that "a prompt increase in heart rate remains the most sensitive indicator of resuscitation efficacy" and that the stethoscope should be the primary means of assessing heart rate (HR). Provision of an accurate and timely HR value is essential if the best care outcomes are to be achieved. Establishing the HR category allows the resuscitator to decide if the HR is >100 bpm (suggests the baby is well or resuscitation is effective), between 60-100bpm (resuscitation required initially focusing on the airway) or <60bpm (requires much more intensive resuscitation which could include CPR). International guidelines recommend assessing the HR every 30 seconds with a stethoscope to track changes and hence efficacy of resuscitation. However, a number of studies demonstrate that newborn healthcare providers estimate the HR category incorrectly in about 1 in 3 cases, potentially resulting in the incorrect management of the baby. There is now strong evidence linking the need for resuscitation and a poor neurodevelopmental outcome in later childhood. Indeed, a number of large cohort studies have demonstrated that even if a baby requires initial resuscitation, and no further need for on-going care, they are at an increased risk of low intelligence quotient in childhood and are less likely to have paid employment or go to University when adults.

More recently electronic stethoscopes (ES) have been used to determine heart rate variability. Several studies have shown that an ES can reliably evaluate the heart rate in adults, but only one recently published study has demonstrated its use in the neonatal patient. The advantage of using an ES over ECG and pulse oximetry is fast acquisition of HR (<5 sec) and ease of application, both attributes are beneficial in the delivery suite scenario. Furthermore, assessment of HR by auscultation (using a stethoscope) is still the primary technique used in many settings.

ECG, an established and accurate method of monitoring HR, is rarely used in the delivery room for a number of reasons including difficulty ensuring adhesion to the skin (the baby is wet/covered in vernix) and skin damage in premature babies caused by stripping of the electrodes. Current ECG systems also require 3 electrodes to be positioned which can delay resuscitation further. To improve HR assessment at birth we aim to tackle this problem through a variety of means. ECG is not routinely used for delivery room resuscitations mainly due to the impracticalities of attaching the electrodes and setting up the system. Current NICU practice is to place the ECG electrodes onto the baby's chest. It is also possible for the electrodes to be placed on the baby's which is a method commonly adopted on the NICU. Preterm babies are routinely delivered into a plastic bags/wraps to minimise heat loss. By pre-placing the ECG electrodes onto the back of the bag/wrap with small conducting holes in, it should be possible to place the baby onto the bag and connect with the ECG electrodes with a routinely used clinical conducting gel. The baby could be placed onto them and time would be saved by not needing to stick the electrodes on individually and utilising the baby's weight to establish the electrode connections. This would avoid the need to place them individually, which is often time consuming and challenging as they don't still well to wet skin, and avoid skin stripping when removed later.

This study will initially assess the accuracy and reliability of an electronic stethoscopes to evaluate heart rate on stable patients on the neonatal unit compared to routine ECG and pulse oximetry measurements. This will allow comparison of the pre placed ECG system in the second phase of the study.

ELIGIBILITY:
Inclusion Criteria:

* All must have written informed consent from the participant's mother
* Phase 1: Any neonate requiring NICU admission and routine monitoring with ECG.
* Phase 2: Preterm infants ≤32 weeks gestation delivered into a plastic bag/wrap

Exclusion Criteria:

* Phase 1: Infants undergoing comfort care (palliative care). Infants deemed too sick, as assessed by the clinical team caring for them, to tolerate additional procedures. This is unusual but would normally include infants who become more unstable with increased handling
* Phase 2: Infants >32 weeks gestation Infants where resuscitation is unlikely to be instigated (eg. known lethal condition)

Max Age: 4 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Phase 1- neonates of any gestation admitted to NICU with routine ECG and pulse oximetry monitoring
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2016-05; Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Heart rate | 10 minutes
  Assessment of accuracy (limits of agreement ±10bpm at 2 standard deviations) and reliability (>90% agreement +/- 10 bpm) of an electronic stethoscope to measure heart rate when compared to ECG.
Reliability of Pre placed ECG leads to measure heart rate | 30 minutes
  Assess of the reliability of pre-placed ECG to measure heart rate at the time of delivery when compared to heart rate assessed by an electronic stethoscope.

SECONDARY OUTCOMES:
Accuracy of Clinical assessment of heart rate using an electronic stethoscope | 30 minutes
  Evaluation of the heart rate by the clinical team when using the electronic stethoscope by subjective counting compared to actual detection of heart rate (computed by software)
Acquisition of video recorded resuscitation of newborns for clinical feedback | 30 minutes
  The resuscitation of the neonate in the delivery room will be recorded to allow alignment of data (i.e. time baby placed in bag, time electronic stethoscope used). This video will be used as a resuscitation training tool for training clinicians.

CONTACTS AND LOCATIONS:
Overall Officials: Don Sharkey, PhD, Principal Investigator — University of Nottingham
Locations (1):
- University of Nottingham NHS Trust, Nottingham, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes